CLINICAL TRIAL: NCT02338973
Title: Pilot Phase I/II Study of the Evaluation of Interferon Gamma-1b Administered Topically for Macular Edema/Intraretinal Schisis Cysts in Rod-Cone Dystrophy (RCD) and Enhanced S-Cone Syndrome (ESCS)
Brief Title: Interferon Gamma-1b Administered Topically for Macular Edema/Intraretinal Schisis Cysts in Rod-Cone Dystrophy (RCD) and Enhanced S-Cone Syndrome (ESCS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150052; 15-EI-0052
Record Dates: First submitted 2015-01-14; First posted 2015-01-15 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2018-07-26

CONDITIONS: Inherited Ophthalmic Diseases; Inherited Retinal Degeneration
Keywords: Macular Edema; Rod-Cone Dystrophy; Inherited Retinal Degeneration; Enhanced S-Cone Syndrome; Interferon Gamma
MeSH Terms: conditions — Macular Edema; Cone-Rod Dystrophies; Enhanced S-Cone Syndrome | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Interferon Gamma-1b (Experimental): Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interventions: Drug: Interferon gamma-1b

INTERVENTIONS:
Drug: Interferon gamma-1b

SUMMARY:
Background:

- People with rod-cone dystrophy (RCD) or enhanced S-cone syndrome (ESCS) have excess fluid under the retina of their eye. This can cause vision loss. The medicine interferon gamma-1b may help people with these diseases.

Objectives:

- To see if interferon gamma-1b eyedrops are safe for people with RCD or ESCS. To see if the medicine can decrease retina fluid and help prevent vision loss.

Eligibility:

- People at least 12 years old with RCD or ESCS. Those with ESCS must have two mutations in the NR2E3 gene.

Design:

* Participants will be screened with medical history, physical exam, eye exam, and blood tests.
* Participants will stay at NIH for 3 days and get the first eyedrops.
* Participants will give themselves 4 study eyedrops 4 times daily for 2 weeks and keep a diary.
* Participants will have 5 outpatient visits over 8 weeks, 2 of which are telephone assessments. They may have:
* Repeats of screening tests.
* Questionnaires.
* Small piece of skin removed.
* Eye exams, including eye dilation and tasks on computer screens.
* Fluorescein angiography. A dye injected into an arm vein will travel to the blood vessels in the eyes. A camera will take pictures.
* Electroretinography. Participants will sit in the dark wearing eyepatches. A small electrode will be taped to the forehead. After 30 minutes, researchers will remove the eyepatches and put in numbing eyedrops and contact lenses. Participants will watch flashing lights.
* Electrooculography. Electrodes will be attached outside of the eyes and eye function will be measured in the dark and the light.
* Participants will have a follow-up visit after 52 weeks.

DETAILED DESCRIPTION:
Objective:

Rod-cone dystrophy (RCD) is a term applied to a number of genetically heterogenous diseases presenting with night vision abnormalities, visual field defects and reduced rod electroretinography responses. Enhanced S-Cone syndrome (ESCS) is a rare autosomal recessive retinal disease with a developmental and a degenerative aspect. Macular cystic changes, often florid and usually resulting in a reduction of central acuity, are frequently associated with both diseases. The reason for this association is not well understood. Acetazolamide (Diamox) and Dorzolamide (Trusopt) have been reported to have variable success in reducing these cystic changes but the effect is frequently inadequate. The objective of this study is to evaluate the safety and potential efficacy of Interferon (IFN) gamma-1b administered topically for macular edema/retinal schisis cysts in RCD and ESCS. Possible disease-related pathophysiologic mechanisms will be explored using induced pluripotent stem cell (iPSC) protocols leading to iPSC-derived retinal pigment epithelium (RPE) and photoreceptor generation.

Study Population:

Up to five participants with RCD with significant macular cystic changes and up to five participants with ESCS with significant macular cystic changes will be enrolled to receive IFN gamma-1b administered topically in one eye. However, up to an additional two participants may be enrolled in order to obtain the five participants in each disease group to be included in the primary analysis if any participants withdraw from the study prior to receiving five days of treatment.

Design:

This is a single-center, prospective, uncontrolled, unmasked pilot Phase I/II study of the safety, tolerability and possible efficacy of IFN gamma-1b in participants with RCD and ESCS and macular cystic changes. One eye of up to five participants with RCD with significant macular cystic changes and up to five participants with ESCS with significant macular cystic changes [evidenced by optical coherence tomography (OCT) >275 microns central macular thickness and/or disruption of foveal contour] will receive topical IFN gamma-1b instilled as drops on the cornea. The initial stage of the study will include two participants from each disease category. Once all four participants have completed the 8-week visit, enrollment will be halted. Safety Adverse Event Review Committee members unaffiliated with the study will review the data as a preliminary assessment of safety and efficacy and to determine whether enrollment should continue. If the committee determines enrollment will continue, three additional participants with RCD and three participants with ESCS will be enrolled. The study will be completed once the final participant has received one year of follow-up.

Outcome Measures:

The primary outcome measure related to the safety and tolerability of IFN gamma-1b administered topically at the prescribed dosage for macular cystic changes in participants with RCD and ESCS will be assessed by the number and severity of adverse events related to the IP and the number of withdrawals at 52 weeks (one year) post-administration. Additional safety of IFN gamma-1b administered topically in participants with RCD and ESCS will be determined from the assessment of retinal function, ocular structure and occurrence of adverse events at all time points. Secondary outcomes include changes in visual function including visual acuity and microperimetry, and retinal imaging with OCT and fluorescein angiography.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant must be 12 years of age or older.
2. Participant (or legal guardian or legal representative) must understand and sign the protocol informed consent.
3. Participant is willing to comply with the study procedures and is expected to be able to return for all study visits.
4. Participant must carry a clinical diagnosis of RCD or ESCS.
5. ESCS participant must have molecular confirmation with two alleles for NR2E3 gene mutations
6. Female participant of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must be willing to undergo pregnancy tests at scheduled study visits.
7. Female participant of childbearing potential, and any male participant able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two reliable methods of contraception while taking the IP and six weeks after completion. Acceptable methods of contraception include:

   * Hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring);
   * Intrauterine device;
   * Barrier methods (diaphragm, condom) with spermicide; or
   * Surgical sterilization (tubal ligation).

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Participant has a history of other ocular disease likely to contribute significantly to visual disruption (e.g., optic neuropathy, glaucoma, uveitis, or other retinal disease).
2. Participant has had diagnosis or treatment of a malignancy (excluding non-melanoma skin cancer) within the previous five years.
3. Participant has received investigational treatment in another clinical study related to an ocular condition in the last six months.
4. Participant is pregnant, lactating, planning to become pregnant (or father a child) during the study follow-up period.
5. Participant is allergic to fluorescein dye.
6. Participant has a systemic condition that, in the opinion of the investigator, would preclude participation in the study (e.g., multiple sclerosis (MS), as IFN gamma may cause MS exacerbations).

Study Eye Eligibility Criteria

A participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

Study Eye Inclusion Criteria

1. The study eye must retain adequate fixation to allow for completion of protocol assessments.
2. The study eye must have macular cystic changes (>275 microns and/or disruption of foveal contour on OCT).

Study Eye Exclusion Criteria

1. The study eye has lens, cornea, or other media opacities that preclude adequate visualization and testing of the retina.
2. The study eye has undergone intraocular surgery within 6 months prior to enrollment.
3. The study eye has a disease that may confound the outcome of the study [e.g., choroidal neovascularization (CNV) in the fovea or parafoveal area].
4. Participant is unwilling to discontinue wearing a contact lens in the study eye during IP administration.

Study Eye Selection Criteria in Cases of Bilateral Disease

RCD and ESCS usually affect both eyes to a similar degree. In case both eyes of a participant meet the study eye eligibility criteria, the following criteria will be used to select the study eye:

* The eye with more intraretinal fluid will be selected as the study eye;
* If both eyes have similar levels of intraretinal fluid, the eye with worse visual acuity will be selected as the study eye;
* If both eyes have the similar levels of intraretinal fluid and visual acuities, the right eye will be selected as the study eye.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01-14; Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wadih Zein, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: People with rod-cone dystrophy (RCD) and enhanced S-cone syndrome (ESCS) were combined as pre-specified in the study protocol
Groups:
- Interferon Gamma-1b: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Period: Overall Study
Arm/Group | Interferon Gamma-1b
Started | 4
Rod-cone Dystrophy (RCD) | 2
Enhanced S-Cone Syndrome (ESCS) | 2
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 45.8 [17 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of IP-related AEs
Description: The number and severity of adverse events related to the investigation product (IP).
Time Frame: Study duration, up to 52 weeks
Measure: Number; unit: adverse events related to IP
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 4
adverse events related to IP
  Severity: Mild | 3
  Severity: Severe | 1

2. Primary Outcome: Number of Participants Who Withdrew
Description: The number of participants who withdrew early.
Time Frame: Study duration, up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Day 1
Description: Change in BCVA from baseline as compared to Day 1 by participant in both study and fellow eyes.
Time Frame: Day 1
Population: BCVA values are presented for Baseline and Day 1 and the change at Day 1 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Baseline in Study Eye; BCVA at Baseline in Fellow Eye; BCVA at Day 1 in Study Eye; BCVA at Day 1 in Fellow Eye; Difference in BCVA at Day 1 From Baseline in Study Eye; Difference in BCVA at Day 1 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Day 1 in Study Eye | BCVA at Day 1 in Fellow Eye | Difference in BCVA at Day 1 From Baseline in Study Eye | Difference in BCVA at Day 1 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 76 | 79 | -1 | -1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 32 | 62 | -7 | 1
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 74 | 70 | 5 | -6
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 18 | 44 | 4 | 2

4. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Day 2
Description: Change in BCVA from baseline as compared to Day 2 by participant in both study and fellow eyes.
Time Frame: Day 2
Population: BCVA values are presented for Baseline and Day 2 and the change at Day 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Day 2 in Study Eye; BCVA at Day 2 in Fellow Eye; Difference in BCVA at Day 2 From Baseline in Study Eye; Difference in BCVA at Day 2 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Day 2 in Study Eye | BCVA at Day 2 in Fellow Eye | Difference in BCVA at Day 2 From Baseline in Study Eye | Difference in BCVA at Day 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 75 | 81 | -2 | 1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 36 | 58 | -3 | -3
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 75 | 69 | 6 | -7
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 21 | 45 | 7 | 3

5. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Day 3
Description: Change in BCVA from baseline as compared to Day 3 by participant in both study and fellow eyes.
Time Frame: Day 3
Population: BCVA values are presented for Baseline and Day 3 and the change at Day 3 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Day 3 in Study Eye; BCVA at Day 3 in Fellow Eye; Difference in BCVA at Day 3 From Baseline in Study Eye; Difference in BCVA at Day 3 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Day 3 in Study Eye | BCVA at Day 3 in Fellow Eye | Difference in BCVA at Day 3 From Baseline in Study Eye | Difference in BCVA at Day 3 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 81 | 78 | 4 | -2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 41 | 61 | 2 | 0
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 74 | 73 | 5 | -3
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 23 | 47 | 9 | 5

6. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Week 2
Description: Change in BCVA from baseline as compared to Week 2 by participant in both study and fellow eyes.
Time Frame: Week 2
Population: BCVA values are presented for Baseline and Week 2 and the change at Week 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Week 2 in Study Eye; BCVA at Week 2 in Fellow Eye; Difference in BCVA at Week 2 From Baseline in Study Eye; Difference in BCVA at Week 2 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Week 2 in Study Eye | BCVA at Week 2 in Fellow Eye | Difference in BCVA at Week 2 From Baseline in Study Eye | Difference in BCVA at Week 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 75 | 78 | -2 | -2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 0 | 66 | -39 | 5
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 66 | 67 | -3 | -9
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 23 | 42 | 9 | 0

7. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Week 5
Description: Change in BCVA from baseline as compared to Week 5 by participant in both study and fellow eyes.
Time Frame: Week 5
Population: BCVA values are presented for Baseline and Week 5 and the change at Week 5 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Week 5 in Study Eye; BCVA at Week 5 in Fellow Eye; Difference in BCVA at Week 5 From Baseline in Study Eye; Difference in BCVA at Week 5 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Week 5 in Study Eye | BCVA at Week 5 in Fellow Eye | Difference in BCVA at Week 5 From Baseline in Study Eye | Difference in BCVA at Week 5 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 71 | 82 | -6 | 2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 0 | 65 | -39 | 4
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 72 | 75 | 3 | -1
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 26 | 45 | 12 | 3

8. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Week 8
Description: Change in BCVA from baseline as compared to Week 8 by participant in both study and fellow eyes.
Time Frame: Week 8
Population: BCVA values are presented for Baseline and Week 8 and the change at Week 8 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Week 8 in Study Eye; BCVA at Week 8 in Fellow Eye; Difference in BCVA at Week 8 From Baseline in Study Eye; Difference in BCVA at Week 8 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Week 8 in Study Eye | BCVA at Week 8 in Fellow Eye | Difference in BCVA at Week 8 From Baseline in Study Eye | Difference in BCVA at Week 8 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 74 | 80 | -3 | 0
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 43 | 65 | 4 | 4
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 72 | 70 | 3 | -6
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 24 | 47 | 10 | 5

9. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline as Compared to Week 52
Description: Change in BCVA from baseline as compared to Week 52 by participant in both study and fellow eyes.
Time Frame: Week 52
Population: BCVA values are presented for Baseline and Week 52 and the change at Week 52 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: letters read
Groups:
- BCVA at Week 52 in Study Eye; BCVA at Week 52 in Fellow Eye; Difference in BCVA at Week 52 From Baseline in Study Eye; Difference in BCVA at Week 52 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | BCVA at Baseline in Study Eye | BCVA at Baseline in Fellow Eye | BCVA at Week 52 in Study Eye | BCVA at Week 52 in Fellow Eye | Difference in BCVA at Week 52 From Baseline in Study Eye | Difference in BCVA at Week 52 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
letters read
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 77 | 80 | 79 | 78 | 2 | -2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 39 | 61 | 47 | 65 | 8 | 4
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 69 | 76 | 65 | 65 | -4 | -11
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 14 | 42 | 20 | 44 | 6 | 2

10. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Day 1
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Day 1 by participant in both study and fellow eyes.
Time Frame: Day 1
Population: Subretinal Fluid Volume values are presented for Baseline and Day 1 and the change at Day 1 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Baseline in Study Eye; Subretinal Fluid Volume at Baseline in Fellow Eye; Subretinal Fluid Volume at Day 1 in Study Eye; Subretinal Fluid Volume at Day1 in Fellow Eye; Difference at Day 1 From Baseline in Study Eye; Difference at Day 1 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Day 1 in Study Eye | Subretinal Fluid Volume at Day1 in Fellow Eye | Difference at Day 1 From Baseline in Study Eye | Difference at Day 1 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 7.35 | 7.35 | 0.1 | 0.25
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 13.95 | 11.25 | -0.2 | 0.05
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 15.15 | 17.2 | -0.95 | -1.35
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 37.7 | 9.2 | 1.4 | -0.05

11. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Day 2
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Day 2 by participant in both study and fellow eyes.
Time Frame: Day 2
Population: Subretinal Fluid Volume values are presented for Baseline and Day 2 and the change at Day 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Day 2 in Study Eye; Subretinal Fluid Volume at Day 2 in Fellow Eye; Difference at Day 2 From Baseline in Study Eye; Difference at Day 2 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Day 2 in Study Eye | Subretinal Fluid Volume at Day 2 in Fellow Eye | Difference at Day 2 From Baseline in Study Eye | Difference at Day 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 7.1 | 7 | -0.15 | -0.1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 14.1 | 10.9 | -0.05 | -0.3
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 15.15 | 15.55 | -0.95 | -3
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 37.3 | 9.05 | 1 | -0.2

12. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Day 3
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Day 3 by participant in both study and fellow eyes.
Time Frame: Day 3
Population: Subretinal Fluid Volume values are presented for Baseline and Day 3 and the change at Day 3 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Day 3 in Study Eye; Subretinal Fluid Volume at Day 3 in Fellow Eye; Difference at Day 3 From Baseline in Study Eye; Difference at Day 3 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Day 3 in Study Eye | Subretinal Fluid Volume at Day 3 in Fellow Eye | Difference at Day 3 From Baseline in Study Eye | Difference at Day 3 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 7.5 | 7.45 | 0.25 | 0.35
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 13.75 | 11.25 | -0.4 | 0.05
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 15.3 | 17 | -0.8 | -1.55
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 35 | 9.1 | -1.3 | -0.15

13. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Week 2
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Week 2 by participant in both study and fellow eyes.
Time Frame: Week 2
Population: Subretinal Fluid Volume values are presented for Baseline and Week 2 and the change at Week 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Week 2 in Study Eye; Subretinal Fluid Volume at Week 2 in Fellow Eye; Difference at Week 2 From Baseline in Study Eye; Difference at Week 2 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Week 2 in Study Eye | Subretinal Fluid Volume at Week 2 in Fellow Eye | Difference at Week 2 From Baseline in Study Eye | Difference at Week 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 7.6 | 7.3 | 0.35 | 0.2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 13.1 | 11 | -1.05 | -0.2
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 14.3 | 17 | -1.8 | -1.55
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 32.5 | 9 | -3.8 | -0.25

14. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Week 5
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Week 5 by participant in both study and fellow eyes.
Time Frame: Week 5
Population: Subretinal Fluid Volume values are presented for Baseline and Week 5 and the change at Week 5 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Week 5 in Study Eye; Subretinal Fluid Volume at Week 5 in Fellow Eye; Difference at Week 5 From Baseline in Study Eye; Difference at Week 5 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Week 5 in Study Eye | Subretinal Fluid Volume at Week 5 in Fellow Eye | Difference at Week 5 From Baseline in Study Eye | Difference at Week 5 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 7.4 | 7.3 | 0.15 | 0.2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 13.9 | 11.2 | -0.25 | 0
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 14 | 15.7 | -2.1 | -2.85
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 29.1 | 9.1 | -7.2 | -0.15

15. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Week 8
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Week 8 by participant in both study and fellow eyes.
Time Frame: Week 8
Population: Subretinal Fluid Volume values are presented for Baseline and Week 8 and the change at Week 8 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Week 8 in Study Eye; Subretinal Fluid Volume at Week 8 in Fellow Eye; Difference at Week 8 From Baseline in Study Eye; Difference at Week 8 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Week 8 in Study Eye | Subretinal Fluid Volume at Week 8 in Fellow Eye | Difference at Week 8 From Baseline in Study Eye | Difference at Week 8 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 7.4 | 7.4 | 0.15 | 0.3
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 13.5 | 10.9 | -0.65 | -0.3
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 13.8 | 17.1 | -2.3 | -1.45
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 27.6 | 9.4 | -8.7 | 0.15

16. Secondary Outcome: Change in Maximum Subretinal Fluid Volume From Baseline as Compared to Week 52
Description: Change in maximum subretinal fluid volume as measured on OCT from baseline as compared to Week 52 by participant in both study and fellow eyes.
Time Frame: Week 52
Population: Subretinal Fluid Volume values are presented for Baseline and Week 52 and the change at Week 52 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: mm^3
Groups:
- Subretinal Fluid Volume at Week 52 in Study Eye; Subretinal Fluid Volume at Week 52 in Fellow Eye; Difference at Week 52 From Baseline in Study Eye; Difference at Week 52 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Subretinal Fluid Volume at Baseline in Study Eye | Subretinal Fluid Volume at Baseline in Fellow Eye | Subretinal Fluid Volume at Week 52 in Study Eye | Subretinal Fluid Volume at Week 52 in Fellow Eye | Difference at Week 52 From Baseline in Study Eye | Difference at Week 52 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
mm^3
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 7.25 | 7.1 | 6.9 | 7 | -0.35 | -0.1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 14.15 | 11.2 | 12.7 | 11.3 | -1.45 | 0.1
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 16.1 | 18.55 | 13.8 | 14.3 | -2.3 | -4.25
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 36.3 | 9.25 | 32.3 | 8.9 | -4 | -0.35

17. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Day 1
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Day 1 by participant in both study and fellow eyes.
Time Frame: Day 1
Population: Central Retinal Thickness values are presented for Baseline and Day 1 and the change at Day 1 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Baseline in Study Eye; Central Retinal Thickness at Baseline in Fellow Eye; Central Retinal Thickness at Day 1 in Study Eye; Central Retinal Thickness at Day 1 in Fellow Eye; Difference at Day 1 From Baseline in Study Eye; Difference at Day 1 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Day 1 in Study Eye | Central Retinal Thickness at Day 1 in Fellow Eye | Difference at Day 1 From Baseline in Study Eye | Difference at Day 1 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 314 | 270.5 | 16.5 | 1.5
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 602 | 298.5 | 5 | 13.5
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 598 | 713.5 | -115 | -70.5
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1394.5 | 232.5 | 1.5 | -9

18. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Day 2
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Day 2 by participant in both study and fellow eyes.
Time Frame: Day 2
Population: Cirrus OCT values are presented for Baseline and Day 2 and the change at Day 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Day 2 in Study Eye; Central Retinal Thickness at Day 2 in Fellow Eye; Difference at Day 2 From Baseline in Study Eye; Difference at Day 2 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Day 2 in Study Eye | Central Retinal Thickness at Day 2 in Fellow Eye | Difference at Day 2 From Baseline in Study Eye | Difference at Day 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 309.5 | 279 | 12 | 10
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 605 | 304.5 | 8 | 19.5
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 613 | 700.5 | -100 | -83.5
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1392.5 | 220 | -0.5 | -21.5

19. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Day 3
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Day 3 by participant in both study and fellow eyes.
Time Frame: Day 3
Population: Cirrus OCT values are presented for Baseline and Day 3 and the change at Day 3 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Day 3 in Study Eye; Central Retinal Thickness at Day 3 in Fellow Eye; Difference at Day 3 From Baseline in Study Eye; Difference at Day 3 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Day 3 in Study Eye | Central Retinal Thickness at Day 3 in Fellow Eye | Difference at Day 3 From Baseline in Study Eye | Difference at Day 3 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 323 | 274 | 25.5 | 5
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 587.5 | 299 | -9.5 | 14
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 621 | 682.5 | -92 | -101.5
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1361.5 | 220 | -31.5 | -21.5

20. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Week 2
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Week 2 by participant in both study and fellow eyes.
Time Frame: Week 2
Population: Cirrus OCT values are presented for Baseline and Week 2 and the change at Week 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Week 2 in Study Eye; Central Retinal Thickness at Week 2 in Fellow Eye; Difference at Week 2 From Baseline in Study Eye; Difference at Week 2 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 2 in Study Eye | Central Retinal Thickness at Week 2 in Fellow Eye | Difference at Week 2 From Baseline in Study Eye | Difference at Week 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 330 | 267 | 32.5 | -2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 534 | 300 | -63 | 15
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 517 | 700 | -196 | -84
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1193 | 208 | -200 | -33.5

21. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Week 5
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Week 5 by participant in both study and fellow eyes.
Time Frame: Week 5
Population: Cirrus OCT values are presented for Baseline and Week 5 and the change at Week 5 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Week 5 in Study Eye; Central Retinal Thickness at Week 5 in Fellow Eye; Difference at Week 5 From Baseline in Study Eye; Difference at Week 5 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 5 in Study Eye | Central Retinal Thickness at Week 5 in Fellow Eye | Difference at Week 5 From Baseline in Study Eye | Difference at Week 5 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 374 | 276 | 76.5 | 7
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 605 | 302 | 8 | 17
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 473 | 580 | -240 | -204
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1083 | 206 | -310 | -35.5

22. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Week 8
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Week 8 by participant in both study and fellow eyes.
Time Frame: Week 8
Population: Cirrus OCT values are presented for Baseline and Week 8 and the change at Week 8 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Week 8 in Study Eye; Central Retinal Thickness at Week 8 in Fellow Eye; Difference at Week 8 From Baseline in Study Eye; Difference at Week 8 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 8 in Study Eye | Central Retinal Thickness at Week 8 in Fellow Eye | Difference at Week 8 From Baseline in Study Eye | Difference at Week 8 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 353 | 276 | 55.5 | 7
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 544 | 224 | -53 | -61
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 456 | 667 | -257 | -117
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1000 | 220 | -393 | -21.5

23. Secondary Outcome: Change in Central Retinal Thickness as Measured on Cirrus OCT From Baseline as Compared to Week 52
Description: Change in central retinal thickness as measured on Cirrus OCT from baseline as compared to Week 52 by participant in both study and fellow eyes.
Time Frame: Week 52
Population: Cirrus OCT values are presented for Baseline and Week 52 and the change at Week 52 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Groups:
- Central Retinal Thickness at Week 52 in Study Eye; Central Retinal Thickness at Week 52 in Fellow Eye; Difference at Week 52 From Baseline in Study Eye; Difference at Week 52 From Baseline in Fellow Eye: Topical interferon (IFN) gamma-1b, 112 µg dose, administered in study eye daily for two weeks
  Interferon gamma-1b
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 52 in Study Eye | Central Retinal Thickness at Week 52 in Fellow Eye | Difference at Week 52 From Baseline in Study Eye | Difference at Week 52 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 297.5 | 269 | 302 | 270 | 4.5 | 1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 597 | 285 | 503 | 307 | -94 | 22
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 713 | 784 | 437 | 457 | -276 | -327
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1393 | 241.5 | 1175 | 197 | -218 | -44.5

24. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Day 1
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Day 1 by participant in both study and fellow eyes.
Time Frame: Day 1
Population: as for outcome 17
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Day 1 in Study Eye | Central Retinal Thickness at Day 1 in Fellow Eye | Difference at Day 1 From Baseline in Study Eye | Difference at Day 1 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 331 | 275 | 24 | -3
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 619 | 319 | 607 | 317 | -12 | -2
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 605 | 703 | -97 | -42
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1418 | 258 | 5 | -2

25. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Day 2
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Day 2 by participant in both study and fellow eyes.
Time Frame: Day 2
Population: Central Retinal Thickness values are presented for Baseline and Day 2 and the change at Day 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Day 2 in Study Eye | Central Retinal Thickness at Day 2 in Fellow Eye | Difference at Day 2 From Baseline in Study Eye | Difference at Day 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 321 | 278 | 14 | 0
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 619 | 319 | 611 | 318 | -8 | -1
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 624 | 682 | -78 | -63
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1427 | 246 | 14 | -14

26. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Day 3
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Day 3 by participant in both study and fellow eyes.
Time Frame: Day 3
Population: Central Retinal Thickness values are presented for Baseline and Day 3 and the change at Day 3 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Day 3 in Study Eye | Central Retinal Thickness at Day 3 in Fellow Eye | Difference at Day 3 From Baseline in Study Eye | Difference at Day 3 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 330 | 277 | 23 | -1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 619 | 319 | 587 | 320 | -32 | 1
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 607 | 656 | -95 | -89
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1393 | 243 | -20 | -17

27. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Week 2
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Week 2 by participant in both study and fellow eyes.
Time Frame: Week 2
Population: Central Retinal Thickness values are presented for Baseline and Week 2 and the change at Week 2 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 2 in Study Eye | Central Retinal Thickness at Week 2 in Fellow Eye | Difference at Week 2 From Baseline in Study Eye | Difference at Week 2 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 333 | 276 | 26 | -2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 619 | 319 | 530 | 317 | -89 | -2
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 552 | 687 | -150 | -58
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1233 | 234 | -180 | -26

28. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Week 5
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Week 5 by participant in both study and fellow eyes.
Time Frame: Week 5
Population: Central Retinal Thickness values are presented for Baseline and Week 5 and the change at Week 5 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 5 in Study Eye | Central Retinal Thickness at Week 5 in Fellow Eye | Difference at Week 5 From Baseline in Study Eye | Difference at Week 5 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 385 | 282 | 78 | 4
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 619 | 319 | 576 | 316 | -43 | -3
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 509 | 591 | -193 | -154
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1089 | 243 | -324 | -17

29. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Week 8
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Week 8 by participant in both study and fellow eyes.
Time Frame: Week 8
Population: Central Retinal Thickness values are presented for Baseline and Week 8 and the change at Week 8 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 8 in Study Eye | Central Retinal Thickness at Week 8 in Fellow Eye | Difference at Week 8 From Baseline in Study Eye | Difference at Week 8 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 370 | 280 | 63 | 2
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 002 | 619 | 319 | 545 | 313 | -74 | -6
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 486 | 657 | -216 | -88
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1020 | 250 | -393 | -10

30. Secondary Outcome: Change in Central Retinal Thickness as Measured on Spectralis OCT From Baseline as Compared to Week 52
Description: Change in central retinal thickness as measured on Spectralis OCT from baseline as compared to Week 52 by participant in both study and fellow eyes.
Time Frame: Week 52
Population: Central Retinal Thickness values are presented for Baseline and Week 52 and the change at Week 52 from Baseline for each participant (study and fellow eye).
Measure: Number; unit: μm
Arm/Group | Central Retinal Thickness at Baseline in Study Eye | Central Retinal Thickness at Baseline in Fellow Eye | Central Retinal Thickness at Week 52 in Study Eye | Central Retinal Thickness at Week 52 in Fellow Eye | Difference at Week 52 From Baseline in Study Eye | Difference at Week 52 From Baseline in Fellow Eye
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 3
μm
  Participant 001: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 001 | 307 | 278 | 309 | 277 | 2 | -1
  Participant 002: number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 0
  Participant 002 | 619 | 319 | 497 |  | -122 |
  Participant 003: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 003 | 702 | 745 | 445 | 472 | -257 | -273
  Participant 004: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
  Participant 004 | 1413 | 260 | 1221 | 233 | -192 | -27

31. Secondary Outcome: Change in Central Visual Field Sensitivity at Day 2 and Week 5 Compared to Baseline.
Description: Change in central visual field sensitivity as measured by microperimetry testing at Day 2 and Week 5 compared to baseline in both study and fellow eyes.
Time Frame: Day 2 and Week 5
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 4
dB
  Day 2 Study Eye | -0.3 (1.6)
  Day 2 Fellow Eye | -1.4 (0.6)
  Week 5 Study Eye | -1.1 (1.1)
  Week 5 Fellow Eye | -1.7 (1.4)

ADVERSE EVENTS:
Time Frame: Up to 52 Weeks
Description: Adverse events were collected on and after the baseline visit, and when investigational product (IP) began.
Arm/Group | Interferon Gamma-1b
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Gamma-1b (N=4)
Visual Acuity Reduced (Eye disorders) | 1 (1) — Decreased vision in OS
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Gamma-1b (N=4)
Ocular Hyperaemia (Eye disorders) | 1 (1) — Mild Redness.
Lacrimation Increased (Eye disorders) | 1 (1) — Tearing
Eye Pruritus (Eye disorders) | 1 (1) — Itching
Cystoid Macular Oedema (Eye disorders) | 1 (1) — Mild Blurring of Vision Due to Worse CME OD
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Abdominal Pain
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back Pain
Retinal Telangiectasia (Eye disorders) | 1 (1) — Idiopathic Juxtafoveal heme
Diabetic Retinopathy (Eye disorders) | 1 (1) — Dot and Blot Heme OS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT02338973/Prot_SAP_000.pdf